CLINICAL TRIAL: NCT05712057
Title: Neurostimulation Enhanced Cognitive Restructuring for Transdiagnostic Emotional Dysregulation: A Component Analysis
Brief Title: Neurostimulation Versus Therapy for Problems With Emotions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00111390; R01MH129302-01A1 (NIH)
Record Dates: First submitted 2023-01-12; First posted 2023-02-03 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Emotion Regulation; Mood Disorders; Stress Disorder; Anxiety Disorders; OCD; Impulse Control Disorder; Eating Disorders; Emotional Dysfunction; Emotional Instability; Emotional Distress; Emotional Maladjustment; Emotional Impulsivity; Obsessive-Compulsive Disorder; Emotion Dysregulation; Borderline Personality Disorder
Keywords: Emotion Dysregulation; Distress Intolerance; Neuromodulation; Neurostimulation; TMS; cognitive restructuring; regulation skills; neuroimaging; Emotion regulation
MeSH Terms: conditions — Emotional Regulation; Mood Disorders; Stress Disorders, Traumatic; Anxiety Disorders; Disruptive, Impulse Control, and Conduct Disorders; Feeding and Eating Disorders; Obsessive-Compulsive Disorder; Borderline Personality Disorder | interventions — Transcranial Magnetic Stimulation; Cognitive Restructuring

STUDY DESIGN:
Intervention Model Description: Group 1 (G1) and 2 (G2) participants will receive training in cognitive restructuring, while Group 3 (G3) participants will receive training in emotional awareness. All participants will undergo negative emotion induction using autobiographical stressors. Depending on group participants could receive one of two types of neurostimulation . Randomization procedures will match subjects on: 1) severity of emotional dysregulation (high/very high), 2) sex at birth, and 3) treatment status (psychotropics/no psychotropics).
Who Masked: Participant, Outcomes Assessor
Masking Description: All participants will engage in a behavioral training session (either cognitive restructuring or emotional awareness training). The clinician who will conduct this behavioral session will be kept blind to thetype of neurostimulation the participant will receive. The neurostimulation technician will be kept blind to the behavioral training that the participant receives. Participants will only be told about the specific type of neurostimulation they receive at the end of the study to protect against different expectations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Cognitive Restructuring + Repetitive Transcranial Magnetic Stimulation (rTMS) (Experimental): Group 1 (G1)- 80 eligible participants will receive training in Cognitive Restructuring (CR). These participants will use CR while receiving rTMS over their individual dlPFC target and will partake in short term and long term follow up testing.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Behavioral: Cognitive Restructuring
- Cognitive Restructuring + scalp electrical stimulation (Active Comparator): Group 2 (G2) - 80 eligible participants will receive training in CR. These participants will use CR while receiving scalp electrical stimulation over their individual dlPFC target and will partake in short term and long term follow up testing.
  Interventions: Device: electrical scalp stimulation; Behavioral: Cognitive Restructuring
- Emotional Awareness Training + Repetitive Transcranial Magnetic Stimulation (rTMS) (Active Comparator): Group 3 (G3) - 80 eligible participants will receive emotional awareness training. These participants will receive rTMS over their individual dlPFC target and will partake in short term and long term follow up testing.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Behavioral: Emotional Awareness Training

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — high frequency rTMS over the right dlPFC
  Other Names: rTMS
  Arms: Cognitive Restructuring + Repetitive Transcranial Magnetic Stimulation (rTMS); Emotional Awareness Training + Repetitive Transcranial Magnetic Stimulation (rTMS)
Device: electrical scalp stimulation — electrical scalp stimulation over the right dlPFC
  Arms: Cognitive Restructuring + scalp electrical stimulation
Behavioral: Cognitive Restructuring — Cognitive restructuring is a cognitive behavioral intervention through which participants learn how to think differently about stressful events in order to feel less emotional arousal.
  Other Names: CR
  Arms: Cognitive Restructuring + Repetitive Transcranial Magnetic Stimulation (rTMS); Cognitive Restructuring + scalp electrical stimulation
Behavioral: Emotional Awareness Training — Emotional awareness training is a behavioral intervention through which participants learn how to identify and evaluate their emotions and the components that make up each emotion.
  Other Names: EAT
  Arms: Emotional Awareness Training + Repetitive Transcranial Magnetic Stimulation (rTMS)

SUMMARY:
The primary goal of this clinical trial is to evaluate the unique neural and behavioral effects of a one-session training combining emotion regulation skills training, with excitatory repetitive transcranial magnetic stimulation (rTMS) over the dorsolateral prefrontal cortex (dlPFC). The secondary aim is to identify key changes in the emotion regulation neural network following the combined intervention versus each of the components alone. The third aim is to explore personalized biomarkers for response to emotion regulation training.

Participants will undergo brain imaging while engaging in an emotional regulation task. Participants will be randomly assigned to learn one of two emotion regulation skills. Participants will be reminded of recent stressors and will undergo different types of neurostimulation, targeted using fMRI (functional MRI) results. Participants who may practice their emotion regulation skills during neurostimulation in a one-time session. Following this training, participants will undergo another fMRI and an exit interview to assess for immediate neural and behavioral changes. Measures of emotion regulation will be assessed at a one week and a one month follow up visit.

DETAILED DESCRIPTION:
Emotional dysregulation constitutes a serious public health problem and novel approaches are needed to effectively address it transdiagnostically. Despite rapid advancements in affective and cognitive neuroscience, there have been few attempts to translate basic findings into novel interventions. In addition, the relevance of different nodes in the emotion regulation network to psychopathology and to successful reduction of emotional arousal is not yet fully understood. Noninvasive neurostimulation, such as repetitive transcranial magnetic stimulation (rTMS), is a powerful tool with which dysfunction can be alleviated temporarily, by modulating neural activation. Therefore, the objective of the current study is to examine immediate neural and behavioral changes following neuromodulation enhanced emotion regulation training for transdiagnostic adults who report difficulties calming down when upset. The central hypothesis is that neurostimulation enhances the acquisition of emotion regulation skills and leads to remediated neural function in the emotion regulation network. The investigators' long-term goal is to develop novel interventions that harness neuroscientific findings to advance behavioral treatments.

The primary aim of this project is to evaluate the unique neural and behavioral effects of a one-session training combining emotion regulation skills with excitatory neurostimulation over the dorsolateral prefrontal cortex (dlPFC). The secondary aim is to identify key changes in the emotion regulation neural network following the combined intervention versus each of the components alone. The third aim is to explore personalized biomarkers for response to emotion regulation training. To achieve these aims, 240 rTMS naïve, community adults who meet criteria for a DSM-5 disorders (excluding if co-occurring anorexia, moderate to severe alcohol and substance use, bipolar I, or psychotic disorders) and who self-report high emotional dysregulation will participate in brain imaging while undergoing an emotional regulation task. Both structural and functional MRI (fMRI) images will be collected. Participants will be randomly assigned to one of three experimental groups that blend neurostimulation and behavioral skills training in different ways. Participants will be reminded of recent autobiographical stressors and will undergo different types of neurostimulation, targeted using fMRI results. Physiological arousal will be monitored throughout the experimental visit. Following this training, 1 week later, participants will undergo another functional scan to assess for immediate neural and behavioral changes. Bio-behavioral measures of emotion regulation will be assessed at this one week visit. The 1-month follow up will occur 1 month after the one week follow-up visit. At this final follow-up visit, participants will also complete an exit interview that assesses acceptability and expectancies as well as a battery of self reports. One final set of bio-behavioral measures of emotion regulation will be completed as well. If successful, the investigators' line of research will provide key mechanistic information to develop a novel transdiagnostic treatment for DSM-5 disorders.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 55
* elevated overall score on Difficulties with Emotion Regulation Scale (DERS total score >=90)
* has been in the same type of psychotherapy (including none) for the last 4 weeks/1mo (*except for current CBT) and is willing to stay on the same regimen throughout the study.
* low self-reported use of cognitive restructuring (ERQ restructuring subscale average score < 4.7)
* meets criteria for at least one mood (including Bipolar II w/o current hypomania), anxiety, stressor, OCD, Impulse Control, ADHD, or eating DSM-5 disorder (except exclusionary diagnoses such as severe anorexia). Note: Both current or partial remission of the disorder will be ok for inclusion into the study.
* verbal agreement to maintain dose of prescribed psychotropic medication (if any) constant throughout the study, provided they are stable on it for the past 4 weeks (except exclusion medication and except if there is a medical emergency requiring changes in medication).
* Naïve to rTMS

Exclusion Criteria:

* current hypomania (Note: Bipolar II w/o current hypomanic episode is ok for inclusion)
* meets diagnostic criteria for current or history of psychotic disorder, or psychotic features,
* meets diagnostic criteria for Bipolar I disorder
* meets diagnostic criteria on SCID5 for current alcohol or substance use disorder (moderate and high severity) or meets past history of severe alcohol use disorder
* unable to read, blind, or deaf, or unwilling to give consent
* non-English speaker,
* verbal IQ < 90 on the North American Adult Reading Test (NART).
* current uncontrolled anorexia or other condition requiring hospitalization
* high risk for suicide defined as either having attempted suicide in past 6 months or reporting current suicidal ideation that includes a method, plan, or intent to die
* current serious medical illness, including current severe migraine headaches
* started/changed psychotropic medications in the prior 4 weeks, or plans to change medication during the study
* history of seizure except those therapeutically induced by ECT (childhood febrile seizures are acceptable and these subjects may be included in the study), history of epilepsy in self or first degree relatives, stroke, brain surgery, head injury, cranial metal implants, known structural brain lesion, devices that may be affected by TMS (pacemaker, medication pump, cochlear implant, implanted brain stimulator), have left elbow/hand/wrist tendonitis
* conditions associated with increased intracranial pressure, space occupying brain lesion, transient ischemic attack, cerebral aneurysm, dementia, Parkinson's or Huntington's disease, multiple sclerosis
* Wellbutrin >300mg per day or on daily stimulant/ADHD medications above the recommended FDA daily recommendations
* use of investigational drug or devices within 4 weeks of screening
* cochlear implants
* Pregnancy
* metal in body that would exclude them from the MRI scan; severe claustrophobia
* is a prisoner or in police custody at time of screening, or has pending court case jeopardizing the participation in the study
* has had TMS in their lifetime
* has had CBT in the past 4 weeks or plans to start therapy during the study
* weighs over 300 pounds (could not fit in MRI scanner)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
High Frequency Heart Rate Variability (HF-HRV) during regulation blocks during the neurostimulation day | Within a month of the initial assessment
  Calculation of physiological data High frequency HRV (HF-HRV) during regulation blocks during the neurostimulation day accounting for baseline controlling for baseline HF-HRV
Time to return to Heart Rate (HR) baseline measured during regulation period | Within a month of the initial assessment
  Following each negative mood induction during the neurostimulation experiment, the time it takes to return baseline HR will be calculated for each of the three regulation periods.
Change in the ventrolateral prefrontal cortex (vlPFC) for the [restructure-flow_negative] contrast | baseline Neuroimaging Scan vs post Neuroimaging scan (1 week follow-up post neurostimulation)
  Change in the maximum activation in the vlPFC from pre-post neuroimaging in the contrast of interest
Change in the dorsomedial prefrontal cortex (dmPFC) for the [restructure-flow_negative] contrast | baseline Neuroimaging Scan, post Neuroimaging Scan (1 week follow-up post neurostimulation)
  Change in the maximum activation in the dmPFC from pre-post neuroimaging in the contrast of interest
Change in the ventromedial prefrontal cortex (vmPFC) for the [restructure-flow_negative] contrast | baseline Neuroimaging Scan, post Neuroimaging Scan (1 week follow-up post neurostimulation)
  Change in the maximum activation in the vmPFC from pre-post neuroimaging in the contrast of interest
Change in the insular cortex for the [restructure-flow_negative] contrast | baseline Neuroimaging Scan, post Neuroimaging Scan (1 week follow-up post neurostimulation)
  Change in the maximum activation in the insula from pre-post neuroimaging in the contrast of interest
Change in dorsolateral prefrontal cortex (dlPFC)-insula connectivity during [restructure - flow_negative] | baseline Neuroimaging Scan, post Neuroimaging Scan (1 week follow-up post neurostimulation)
  Using Generalized Psychophysiological Interaction (gPPI) analysis the difference in dlPFC-insula connectivity pre-post neuromaging
Change in dorsolateral prefrontal cortex (dlPFC)-amygdala connectivity during [restructure - flow_negative] | baseline Neuroimaging Scan, post Neuroimaging Scan (1 week follow-up post neurostimulation)
  Using Generalized Psychophysiological Interaction (gPPI) analysis the difference in dlPFC-amygdala connectivity pre-post neuromaging

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS) self-report change | Baseline, 1 week follow-up after neurostimulation, 1 month follow-up
  Change in self-reported DERS will be investigated immediately after the followup neuroimaging session and one month after training. DERS inclusion for study is a score of 90 or higher. Min-Max score ranges from 36-180 (with higher scores signifying more difficulties with emotion regulation)
Emotion Regulation Questionnaire (ERQ) self-report change | Baseline, 1 week follow-up after neurostimulation, 1 month follow-up
  Change in Self-reported use of Cognitive Restructuring (CR) as measured with the Emotion Regulation Questionnaire (ERQ) one week and one month after training. We will also examine pre-post changes in ERQ-Reappraisal scale using a similar growth model approach, accounting for severity of psychopathology and baseline. The ERQ is a 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal (6 scale items) and (2) Expressive Suppression (4 scale items). Scores for the 2 scales are reported the average score of the total items in that scale. The lower the average score on the reappraisal scale the more problems with regulating emotions.
Change in the dlPFC for the [restructure - flow_negative] contrast | baseline Neuroimaging scan, post Neuroimaging Scan (1 week follow-up neurostimulation)
  Change in the maximum activation in the dlPFC from pre-post neuroimaging in the contrast of interest
Change in the amygdala for the [restructure - flow_negative] contrast | baseline Neuroimaging scan, post Neuroimaging Scan (1 week follow-up neurostimulation)
  Change in the maximum activation in the amygdala from pre-post neuroimaging in the contrast of interest
Outcome Questionnaire (OQ-45) self-report change | Baseline, 1 week follow-up after neurostimulation, 1 month follow-up
  Change in self-reported psychopathology as measured by the OQ-45 one week and one month after training. The Outcome Questionnaire-45 (OQ-45) is a 45-item self-report measure used to track severity of psychopathology throughout treatment. It consists of subscales that identify three types of problems that lead to general stress: psychological symptoms, interpersonal conflicts, and problems with social roles. Items are rated on a Likert scale ranging from 0 (never) to 4 (almost always). Scores range from 0 to 180. Higher scores indicate higher psychopathological distress than lower scores.
Cognitive Skills Questionnaire (CSQ) self-report change | Baseline, 1 week follow-up after neurostimulation, 1 month follow-up
  Change in self-reported use of cognitive skills as measured by the CSQ one week and one month after training. The CSQ is the Unified Protocol Cognitive Skills Questionnaire (UPCSQ; unpublished) that contains 8 items that ranges from "1" Never to "5" Always or When Needed with higher scores indicating more use of tools or skills than lower scores. Scores range from 8 to 40 (highest skill use).
Self Efficacy with Emotion Regulation (PROMIS-SEME) | Baseline, 1 week follow-up after neurostimulation, 1 month follow-up
  Change in effective regulation as measured by PROMIS-SEME from baseline to follow up. PROMIS Self-Efficacy for Managing Emotions measures one's confidence to manage emotions such as anxiety, helplessness, and discouragement on a scale of 1 "not at all confident" to 5 "I am very confident." There are total of 25 items with a score ranging from 25 to 125. Higher scores indicate higher confidence in the ability to use emotion regulation skills. Scores are then reported using the PROMIS manual for T-scores.
Change in subjective units of distress (SUDS) | Neurostimulation visit (which will occur within a month of the initial assessment)
  SUDS measured after baseline, stressor and every three minutes during regulation, including at the end of regulation during the neurostimulation experiment
HF-HRV during regulation block at follow up | one week follow-up, 1 month follow-up
  Change in HF-HRV mean during regulation block of stressor task at neurostimulation visit at follow-up
Time to return to HR baseline measured during regulation period at follow up | one week follow-up, 1 month follow-up
  time it takes to return baseline HR will be calculated during the behavioral stressor computer task at follow up

OTHER OUTCOMES:
Change in vmPFC-insula connectivity during [restructure - flow_negative] | baseline Neuroimaging scan, post Neuroimaging Scan (1 week follow-up neurostimulation)
  Using Generalized Psychophysiological Interaction (gPPI) analysis the difference in vmPFC-insula connectivity pre-post neuromaging
Cognitive flexibility inventory (CFI) and cognitive control and flexibility inventory (CCFI) | Baseline
  CFI and CCFI total scores will be used as a moderator of outcomes. The CFI is a 20-item self-report measure to monitor how often individuals engaged in cognitive behavioral thought challenging interventions. Scores consist of a total CFI score and two subscale scores. The total score ranges between 20 and 140, where higher scores indicate more cognitive flexibility. The CCFI is an 18 item measure that assesses an individual's perceived ability to exhibit control over their thoughts and behavior in a stressful situation on a scale of "1" Strongly Disagree to "7" Strongly agree with a range from 18-126. Higher scores on the CCFQ were most strongly related to greater cognitive reappraisal as well as less perseverative thinking and rumination.
Wisconsin Card Sorting Task | Baseline
  Behavioral measurement of cognitive flexibility achieved with the wisconsin card sort will be used as a moderator of outcomes
Affect Intensity Measure (AIM) | Baseline
  AIM total score will be used as a moderator of outcomes. The AIM is a 40-item questionnaire designed to measure the characteristic strength or weakness with which one experiences emotion where participants rate from "1" Never to "6" Always with higher scores meaning higher emotion intensity than lower scores.

CONTACTS AND LOCATIONS:
Overall Officials: Andrada D Neacsiu, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be submitted to the National Institute of Mental Health Data Archive (NDA) at the National Institutes of Health (NIH). NDA is a large database where deidentified study data from many NIH studies are stored and managed. NDA is run by the National Institute of Mental Health (NIMH) that allows researchers studying mental illness and brain science to collect and share deidentified information with each other. When the study team sends the data to the NIMH, they will do this through a password secure system where participants are identified by a specific GUID which is a unique # representing 1 specific person in the nation.
  NIMH will also report to Congress and on its website about the different studies using NDA data. Participants can decide that they do not want to share their information to NDA.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Either on a rolling basis over the life of the grant/project per NDA's sharing calendar. Otherwise, within 6 months of completing participant data collection or very soon after publication of primary aims.
Access Criteria: Users with NDA credentials must submit Data Access Requests for one NDA Permission Group at a time. Each DAR requires an NDA Data Use Certification (DUC) signed by the lead recipient and an authorized Signing Official from the recipient's research institution. All recipients on a Data Access Request/Data Use Certification must be affiliated with the lead recipient's research institution. If the Lead Recipient on a DUC changes institutions, they may identify another Recipient on the DUC as a replacement.
  Data Access Requests for a given NDA Permission Group are reviewed by one NIH-staffed Data Access Committee (DAC).
  Detailed information about NDA permission groups is maintained at https://nda.nih.gov/nda/about-us.html.
  When approved to access, teams have access to query and download all data available using the NDA Query Tool and NDA download tools.